CLINICAL TRIAL: NCT06380829
Title: Psychometric Properties of the Self-Care Assessment Scale for 3-6 Year Old Children With Cerebral Palsy-Parent Form: Turkish Validity and Reliability Study
Brief Title: Psychometric Properties of the Self-Care Assessment Scale for 3-6 Year Old Children With Cerebral Palsy-Parent Form
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Bircan Kahraman Berberoglu, research asistant, Aydin Adnan Menderes University
Other Study IDs: Adnan Menderes
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy; Self Care
MeSH Terms: conditions — Cerebral Palsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Self-Care Assessment Scale for Children with CP aged 3-6 years - Parent Form (SPÇÖS-EF): A draft scale named SPÇÖS-EF was prepared by the researchers, using the literature, to determine the self-care status of children with cerebral palsy aged 3-6.

SUMMARY:
This study is a methodological study to develop the self-care assessment scale-parent form of children with CP aged 3-6 years and test its validity and reliability.

Q1. Is the Self-Care Assessment Scale for 3- to 6-year-old Children with CP a valid scale? Q2. Is the Self-Care Assessment Scale for 3- to 6-year-old Children with CP a reliable scale?

DETAILED DESCRIPTION:
This methodological research was conducted with the parents of 127 children with cerebral palsy aged 3-6 years old who were receiving education in special education and rehabilitation centers. Data were collected using the Child-Parent Information Form and the Self-Care Assessment Scale for Children with CP aged 3-6 years Parent Form (SPÇÖRS-EF). Descriptive statistics, Kruskal-Wallis, Cronbach alpha, test-retest, Kaiser-Meyer-Olkin (KMO) test, Bartlett test, explanatory factor analysis and confirmatory factor analysis were used to analyze the data. The research was conducted with the parents of children aged 3-6 years old with cerebral palsy who came to nine special education and rehabilitation centers in four provinces in western Turkey to receive physical therapy between June 5 and December 5, 2023. The sample of the study was calculated by taking at least five times the total number of items in the scale (25 items*5=125, n=125). Non-probability random sampling method was used in sample selection. The research was completed with the participation of 127 parents. According to post hoc power analysis, this sample size was confirmed to be sufficient for 97% power (with a medium effect size d = 0.3 and α = 0.05 type I error). Criteria for inclusion in the study; The children were between the ages of 3-6 (36-72 months), lived with their parents, and the parents were at least literate and able to speak and understand Turkish. This study was conducted in accordance with the Helsinki Declaration and was approved by Aydın Adnan Menderes University Nursing Faculty Non-Interventional Ethics Committee (Date: 27.04.2023, Number: 2023/350). Verbal consent of the participants was obtained. Written permission was obtained from the special education and rehabilitation centers where the research was conducted.

ELIGIBILITY:
Inclusion Criteria:

Being between 3-6 years old (36-72 months) living with their parents

Exclusion Criteria:

be at least literate He/she was able to speak and understand Turkish.

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Children with CP between the ages of 3-6
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
To asses Turkish validity and reliability of Self-Care Assessment Scale for Children with CP aged 3-6 years | six month from the beginning of the study
  This study is a methodological study to develop the self-care assessment scale-parent form of children with CP aged 3-6 years and test its validity and reliability. The scale includes 24 items to question the child's self-care skills, such as independent nutrition, eating, being able to express himself while meeting his basic needs, toileting, dressing, washing hands and face, brushing teeth, cleaning his nose and expressing himself when he is sleepy, in accordance with his age. The scale is a 5-point Likert type, and each item is scored between 1-5, from "Always (independent)" to "Never (completely dependent)". In the scale, the 4th, 8th, 17th, 23rd scale items are reversed to obtain the total scale score. A minimum of 24 and a maximum of 120 points can be obtained from the scale. A high score from the scale indicates that the child with CP has good self-care skills.

CONTACTS AND LOCATIONS:
Overall Officials: BIRCAN KAHRAMAN BERBEROĞLU, PHD, Principal Investigator — Aydın Adnan Menderes Univercity
Locations (1):
- Bircan Kahraman Berberoğlu, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahraman Berberoglu B, Calisir H. The effect of structured supportive approach based on Kolcaba's comfort theory applied to parents of children with cerebral palsy on child's comfort, quality of life, and parent's self-efficacy: A randomised controlled trial. J Pediatr Nurs. 2024 Mar-Apr;75:e65-e74. doi: 10.1016/j.pedn.2023.12.032. Epub 2024 Jan 20. PMID 38246818